CLINICAL TRIAL: NCT06614673
Title: Cancer Literacy as An Essential factoR for Lifestyle behaviOr Changes: An Observational and Interventional Study
Acronym: CLARO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Collaborators: University of Music, Drama, and Media Hannover (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CLARO main stuy
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-02

CONDITIONS: Cancer Prevention
Keywords: Cancer; Cancer Literacy; Informational Intervention; Health Communication
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Non-Narrative Text (Experimental): A short text, consisting of 504 words, that addresses the preventability of cancer cases. It highlights the impact of lifestyle factors such as smoking, unhealthy diet, obesity, and physical inactivity, which contribute to approximately 40% of cancer cases. The text also provides recommendations for reducing the risk of cancer through behavioral changes in these areas, with a particular emphasis on nutrition and physical activity. The text was developed based on the Protection Motivation Theory.
  Interventions: Other: text in non-narrative form
- Narrative Text (Experimental): The narrative text contains the same information as the non-narrative text, but it is presented as a story. It is slightly longer at 737 words and features a main character and two work colleagues sharing their personal experiences about nutrition and physical activity.
  Interventions: Other: text in narrative form
- Non-Narrative Animation (Experimental): The animation with a total duration of 3:35 min is based on the text in non-narrative form and aims to be as fully comparable as possible.
  Interventions: Other: animated video in non-narrative form
- Narrative Animation (Experimental): The animaion (4:04 min) is based on the text in narrative form and aims to be as fully comparable as possible.
  Interventions: Other: animated video in narrative form
- Control Group (No Intervention): After completing all the questionnaires (i.e. after completing participation in the study), the control group will be given the opportunity to view all the information material that was created.

INTERVENTIONS:
Other: text in non-narrative form — Participants will be asked to read a text and complete questionnaires
  Arms: Non-Narrative Text
Other: text in narrative form — Participants will be asked to read a text and complete questionnaires
  Arms: Narrative Text
Other: animated video in non-narrative form — Participants will be asked to watch a video and complete questionnaires
  Arms: Non-Narrative Animation
Other: animated video in narrative form — Participants will be asked to watch a video and complete questionnaires
  Arms: Narrative Animation

SUMMARY:
The CLARO study aims to examine the most effective way to design information materials that can strengthen optimistic beliefs about cancer prevention and improve cancer literacy indirectly. Around 5,800 participants from the Stuttgart region in Germany will be contacted by postal mail and invited to take part in an online survey using the LimeSurvey®-System. Four different types of information materials, tested in a pilot study (2x2-design: text or animation-based / narrative or non-narrative), will be included in the survey. Participants will be randomly assigned to one of the four interventions or to a control group that will not receive any intervention (the control group will have access to all information materials after having completed the whole questionnaire). As an incentive, participants will receive 10€ via bank transfer upon completing the survey.

DETAILED DESCRIPTION:
The online survey can be accessed through a unique link or QR code and is compatible with various electronic devices such as PCs, tablets, and smartphones. Reminders will be sent after one month and two months. Participants can also request a paper questionnaire if needed. We will make an effort to contact more people from districts with lower socioeconomic status. Furthermore, the study cover letter will disclose that all study participants will receive ten euros if they provide their bank details after completion of the study questionnaires. Participants will be redirected via a link to another LimeSurvey for this purpose.

The online questionnaire will be divided into two parts. The first part, which will assess sociodemographic information, questions on cancer literacy, and more, will take about 10 minutes. Subsequently, participants will be randomly assigned to one of the four intervention groups or to a control group. Reading or viewing the information materials will take about 5 minutes. In the second part of the questionnaire, participants will evaluate the information materials, assess intentions for health behaviors, and have access to further information materials (approximately 5 minutes). The control group will have access to all information materials after having completed the whole questionnaire.

The primary aims of the observational part of the study are, first, to assess levels of cancer literacy in a representative German population, including all four cancer literacy domains (i.e., access, understand, appraise, apply). Second, this study part aims to identify sociodemographic groups (e.g., defined by age, sex, sociodemographic background, educational level) showing significantly lower levels of cancer literacy. As a secondary aim, the observational part of the study determines levels of cancer prevention behaviors in Germany (i.e., smoking status, diet, alcohol consumption, and physical activity).

The primary aim of the interventional part of the study is to assess the effects of different health communication strategies (i.e., text or animation in non-narrative or narrative style) on the primary outcome of cancer prevention beliefs. The secondary aim is to examine health communication strategies in their effect on secondary outcomes, i.e., intention for cancer prevention behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 70 years old
* Being able to speak and understand german

Exclusion Criteria:

* Not being able and willing to provide informed consent and complete questionnaires

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1422 (Actual)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Awareness for cancer risk factors | 5 Minutes
  Sixteen cancer risk factors from the Cancer Awareness Measure (CAM), will be assessed. Additionally, the Mythical Causes Scale of the Cancer Awareness Measure (CAM-MYCS) will be included which asks for 11 factors commonly believed to cause cancer, although there is no scientific evidence (e.g., drinking from plastic bottles). recommendations, will be assessed.
Knowledge of the European Code Against Cancer recommendations | 2 Minutes
  Cancer risk factors, that are not part of the CAM, but mentioned in the ECAC4 recommendations, will be assessed.
Cancer prevention beliefs | 1 Minute
  i.e., beliefs how much cancer development is controllable by own behavior choices, will be assessed by asking for agreement with three statements that have been used in previous studies: "It seems like everything causes cancer," "There's not much you can do to lower your chances of getting cancer," and "There are so many recommendations about preventing cancer, it's hard to know which ones to follow".It has been argued that the third item is actually not targeting cancer prevention beliefs, but cancer information overload, which is why it also appears in the Cancer Information Overload Scale.
Information retrieval | 5 Minutes
  Information retrieval will be assessed with three items of the CAM, assessing (1) whether information on cancer prevention has ever been looked for, if yes: (2) sources of information (8 answer options), and (3) features of information sources that played a role for the decision to use information (11 answer options; if no: (2) sources of information they would use (8 answer options), and (3) features of information sources that would play a role for the decision to use information (11 answer options). Additionally, we will assess the perception of being overwhelmed by too much information on cancer prevention using the second item of the cancer prevention beliefs. Active information search will be objectively measured by offering participants informational materials on different prevention behaviors and measuring interest in downloads within the survey.
Japanese Cancer Intelligence Quotient | 1 Minute
  Two selected items from the Japanese Cancer Intelligence Quotient (JCIQ) will additionally assess participants' capability to appraise and apply informations regarding cancer risk.

SECONDARY OUTCOMES:
Health Literacy | 3 Minutes
  We will assess Health Literacy using the short form of the European Health Literacy Survey HLS-Q12 , addressing self-reported competencies in accessing, understanding, appraising, and applying the information in decisions-making in healthcare, disease prevention, and health promotion.
Sociodemographic variables | 3 Minutes
  age, sex, income,education, professional activity, migration background
Personal variables | 2 Minutes
  cancer history, friends or family with cancer

CONTACTS AND LOCATIONS:
Overall Officials: Karen Steindorf, Prof. Dr., Principal Investigator — German Cancer Research Center; Alexander Haussmann, Dr., Principal Investigator — German Cancer Research Center; Florian Herbolsheimer, Dr., Principal Investigator — German Cancer Research Center
Locations (1):
- German Cancer Research Center, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No